CLINICAL TRIAL: NCT05547126
Title: Comparing Different Montages of Transcranial Direct Current Stimulation Combined With Dual-task Training on EEG Microstates A Proof-of-concept Study
Brief Title: Comparing Different Montages of tDCS Combined With Dual-task Training on EEG Microstates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Suellen Marinho Andrade, Federal University of Paraíba, Federal University of Paraíba
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: tDCS+Dual-tasktraining_Stroke
Record Dates: First submitted 2022-08-18; First posted 2022-09-21 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Stroke
Keywords: Transcranial direct current stimulation; Stroke; Dual-task training; EEG
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Anodal tDCS + dual-task training (Active Comparator): The anodic electrode (5x5 cm) will be applied to the primary motor area (C3/C4) ipsilateral to the lesion and the reference electrode (6x9 cm) to the deltoid muscle region.
  Simultaneously with the tDCS sessions, participants will be submitted a protocol based on motor and cognitive dual-task training. The dual-task training will have a total duration of 20 minutes in each session.
  Interventions: Device: Transcranial direct current stimulation
- tDCS dualsite + dual-task training (Active Comparator): Two active electrodes (5x5 cm) will be used, which will be positioned over the primary motor area (C3/C4) and over the dorsolateral prefrontal cortex (F3 or F4) in the ipsilateral hemisphere. For this stimulation modality, two active electrodes (anodic) and a reference electrode (6x9 cm) will be used on the deltoid muscle region.
  Simultaneously with the tDCS sessions, participants will be submitted a protocol based on motor and cognitive dual-task training. The dual-task training will have a total duration of 20 minutes in each session.
  Interventions: Device: Transcranial direct current stimulation
- tDCS sham + dual-task training (Placebo Comparator): Two electrodes will be used, which will be positioned over the primary motor area (C3/C4) and a reference electrode (6x9 cm) will be used on the deltoid muscle region, however the device will be configured in sham mode.
  Simultaneously with the tDCS sessions, participants will be submitted a protocol based on motor and cognitive dual-task training. The dual-task training will have a total duration of 20 minutes in each session.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — It is currently known that Transcranial Direct Current Stimulation (tDCS) can modulate cortical activity, being considered an important resource in the treatment of sequelae resulting from stroke.
  Cognitive motor dual-task training (CMDT) is a type of cognitive rehabilitation training at the same time as exercise rehabilitation therapy.
  Other Names: tDCS; Dual-task training

SUMMARY:
This study investigates whether electroencephalographic (EEG) measures of functional connectivity of the target network are associated with the response to different sets of transcranial direct current stimulation combined with dual-task training in post-stroke patients.

DETAILED DESCRIPTION:
The present study seeks to compare the effects of conventional anodic tDCS (M1) with double-site/dual-site anodic tDCS (M1 + DLPFC) and simulated tDCS on functional connectivity, as assessed by EEG, in patients after staged stroke. chronic. The study is a randomized, double-blind, placebo-controlled, crossover clinical trial. Participants will be submitted to three sessions, each session consisting of a different condition, namely: anodic tDCS - participants who will receive real current over the primary motor area; Dualsite tDCS - participants who will receive real current over the primary motor area and over the dorsolateral prefrontal area (DLPFC) and simulated tDCS - participants who will receive simulated stimulation. Participants will receive 3 tDCS sessions, lasting 20 minutes, associated with a physical therapy protocol based on dual motor and cognitive tasks, on alternate days (3 times a week). On each intervention day, pre and post-intervention assessments will be carried out, the evaluated outcomes will be: functional connectivity (EEG), functional mobility (Timed Up and Go) and executive functions (Trail-making Test A and B, the Clock Drawing Test and Phonemic Verbal Fluency Test). Statistical performance will be performed using SPSS software (Version 20.0) and MATLAB 9.20 with a significance level of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Post-stroke participants for more than 6 months
* Individuals over 18 years of age;
* Both sexes;
* Patients with mild to moderate degree of injury severity (NIHHS <17 points)

Exclusion Criteria:

* Patients with other associated pathologies that can influence motor activity (example: traumatic brain injury, brain tumor);
* Habitual use of drugs or alcohol;
* Use of drugs that modulate the activity of the Central Nervous System;
* Gestation;
* Use of metallic / electronic implants and / or cardiac pacemakers;
* Participants unable to communicate verbally;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Microstates EEG | The evaluations will be carried out in pre-intervention
  EEG data were processed according to the following steps and parameters: (1) downsampled to 256 Hz; (2) high-pass filter at 2 Hz and low-pass at 20 Hz; (3) visual inspection and artifact removal; (4) correction of eye movement using the independent component analysis; and (5) segmentation into two-second epochs with 10% overlap. The choice for the 2-20 Hz range frequency band. Data were submitted to processing: determination of global field power; clustering using k-means of topographic maps of global field power peaks; determination of the optimal number of topographic maps using a predetermined criterion of the four classic maps (A, B, C, and D); application of the topographic maps to the EEG signal using spatial correlation; and classification of EEG continuous data according to the topographic map with the most correlated sections. We calculated and extracted the global explained variance, coverage, occurrence, and duration from each topography.
Functional connectivity | Immediately after the intervention
  EEG data were processed according to the following steps and parameters: (1) downsampled to 256 Hz; (2) high-pass filter at 2 Hz and low-pass at 20 Hz; (3) visual inspection and artifact removal; (4) correction of eye movement using the independent component analysis; and (5) segmentation into two-second epochs with 10% overlap. The choice for the 2-20 Hz range frequency band. Data were submitted to processing: determination of global field power; clustering using k-means of topographic maps of global field power peaks; determination of the optimal number of topographic maps using a predetermined criterion of the four classic maps (A, B, C, and D); application of the topographic maps to the EEG signal using spatial correlation; and classification of EEG continuous data according to the topographic map with the most correlated sections. We calculated and extracted the global explained variance, coverage, occurrence, and duration from each topography.

SECONDARY OUTCOMES:
Timed up and Go test | The evaluations will be carried out in pre-intervention
  Timed up and Go test
Timed up and Go test | Immediately after the intervention
  Timed up and Go test
Executive Functions I | The evaluations will be carried out in pre-intervention
  Trial-making Test A and B
Executive Functions I | Immediately after the intervention
  Trial-making Test A and B
Executive Functions II | The evaluations will be carried out in pre-intervention
  the Clock Drawing Test
Executive Functions II | Immediately after the intervention
  the Clock Drawing Test
Executive Functions III | The evaluations will be carried out in pre-intervention
  Phonemic Verbal Fluency Test
Executive Functions III | Immediately after the intervention
  Phonemic Verbal Fluency Test

CONTACTS AND LOCATIONS:
Overall Officials: Suellen Andrade, Principal Investigator — Federal University of Paraíba
Locations (1):
- Federal University of Paraíba,Department of Psychology, João Pessoa, Paraíba, Brazil